CLINICAL TRIAL: NCT03192358
Title: Physiological Flow of Liquids Used in Dysphagia Management
Brief Title: Physiological Flow of Liquids Used in Dysphagia Management (Neuro)
Status: Completed | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Collaborators: University of Florida (Other); National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Sponsor
Other Study IDs: 17-5421; 5R01DC011020-05 (NIH); CAPCR 17-5421 (NIH_Neuro) (Other: University Health Network Research Ethics Board); IRB201701608 (Other: University of Florida Institutional Review Board)
Record Dates: First submitted 2017-06-12; First posted 2017-06-20 (Actual); Results first posted 2022-07-14 (Actual); Last update posted 2022-09-15 (Actual); Status verified 2021-03

CONDITIONS: Amyotrophic Lateral Sclerosis; Parkinson Disease; Dysphagia
Keywords: Thickened Liquids; Dysphagia Management; Videofluoroscopy; Swallowing Physiology
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Parkinson Disease; Deglutition Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Amyotrophic Lateral Sclerosis: We will be recruiting individuals with confirmed or probably ALS, who experience speech or swallowing problems, to attend one data collection session. All participants will undergo the same protocol, including a Videofluoroscopic Swallowing Examination, and Tongue Strength Measurement.
  Interventions: Diagnostic Test: Videofluoroscopic Swallowing Examination; Other: Tongue Strength Measurement
- Parkinson's Disease: We will be recruiting individuals with a diagnosis of Parkinson's disease, who experience speech or swallowing problems, to attend one data collection session. All participants will undergo the same protocol, including a Videofluoroscopic Swallowing Examination, and Tongue Strength Measurement.
  Interventions: Diagnostic Test: Videofluoroscopic Swallowing Examination; Other: Tongue Strength Measurement

INTERVENTIONS:
Diagnostic Test: Videofluoroscopic Swallowing Examination — During the videofluoroscopy, subjects will take up to 21 sips of liquid, ranging in thickness from thin (like water), to extremely-thick (like pudding or custard). The liquids will be mixed with E-Z-Paque barium sulfate, to allow it to be visible on the x-ray.
Other: Tongue Strength Measurement — We will measure tongue strength using a tongue pressure measurement system called the Iowa Oral Performance Instrument (IOPI). A small disposable bulb filled with air will be placed in the mouth, just behind the front teeth. Participants will be asked to press their tongue upwards against the bulb as hard as they can, three (3) times at the front of the tongue and three (3) times at the back of the tongue (i.e., total of six (6) maximum isometric tongue presses). Participants will also be asked to swallow their saliva with the bulb placed in their mouth, three (3) times.
  Tongue pressure measurement will be completed twice in the data collection session - once at the beginning, and once at the end (following the videofluoroscopy).

SUMMARY:
For individuals with neurodegenerative conditions, such as Amyotrophic Lateral Sclerosis and Parkinson disease, swallowing impairment (i.e., dysphagia) is a common and serious symptom. Dysphagia places the affected individual at risk for secondary health consequences, including malnutrition and aspiration pneumonia, and negatively affects quality of life.

Thickened liquids are commonly recommended for individuals with dysphagia, as they flow more slowly and reduce the risk of entry into the airway. However, there is limited understanding about how changes in liquid thickness modulate swallowing physiology in individuals with neurodegenerative conditions, and previous reports have shown that increased liquid thickness may contribute to the accumulation of residue in the throat.

The purpose of this study is to explore swallowing physiology and function in individuals with neurodegenerative conditions, across five levels of liquid thickness (thin, slightly-thick, mildly-thick, moderately-thick, and extremely-thick), and to identify boundaries of "optimal liquid thickness", which maintain airway safety, without contributing to the accumulation of significant residue. Results from this study will help guide the clinical recommendations for thickened liquids in dysphagia management.

DETAILED DESCRIPTION:
This observational research study will measure swallowing function in individuals with Amyotrophic Lateral Sclerosis or Parkinson's disease. The aims of this study are to (1) identify parameters of swallowing physiology that are associated with impaired swallowing safety and efficiency, and (2) explore how liquid thickness influences swallowing function.

Participation in this research study involves a single appointment at the University of Florida Swallowing Systems Core laboratory located at Shands Hospital, Gainesville. The appointment will last approximately 1 hour, and will involve tasks to measure tongue-strength, and a dynamic swallowing x-ray (known as videofluoroscopy) to evaluate swallowing function. A selection of demographic information (e.g., age, onset of symptoms) will also be recorded.

To measure tongue strength, participants will be given a disposable air-filled bulb and asked to perform a series of tongue presses, and swallow their saliva. Next, during the videofluoroscopy, participants will take sips of various liquids ranging in thickness from thin (like water), to extremely-thick (similar to the consistency of pudding or yogurt). The liquids will be mixed with a safe substance called barium, to make them visible on x-ray images. After the videofluoroscopy has been completed, each participant will have their tongue strength measured again, which will conclude their participation in the study.

Swallowing physiology will be measured from the videofluoroscopy images, post-hoc, by an experienced team of blinded raters.

ELIGIBILITY:
Inclusion Criteria:

* Adults (18+) with a confirmed diagnosis of Amyotrophic Lateral Sclerosis (ALS) or Parkinson's disease (PD)

Exclusion Criteria:

* People with a prior medical history of stroke
* People with a prior medical history of acquired brain injury
* People with a prior medical history of spinal or spinal cord injury
* People with a prior medical history of cancer or surgery in the head and neck region
* People who have had radiation to the head and neck for cancer
* People who have a prior history of swallowing problems (e.g., from childhood, medical complication)
* People with significant breathing difficulties (e.g., rely on mechanical ventilation)
* People who rely solely on tube-feeding for all meals and nutrition
* People who have Type I (insulin-dependent) Diabetes
* Women who are pregnant
* People who have allergies to barium, potato starch, corn starch, xanthan gum, milk products, latex or dental glue

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with ALS will be recruited from the multidisciplinary ALS clinics at the University of Florida during regularly scheduled care visits. Participants with Parkinson's disease will be recruited from the University of Florida Center for Movement Disorders.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Catriona M Steele, PhD, Principal Investigator — University Health Network - Toronto Rehabilitation Institute; Emily K Plowman, PhD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pearson WG Jr, Molfenter SM, Smith ZM, Steele CM. Image-based measurement of post-swallow residue: the normalized residue ratio scale. Dysphagia. 2013 Jun;28(2):167-77. doi: 10.1007/s00455-012-9426-9. Epub 2012 Oct 23. PMID 23089830
- [Background] Rosenbek JC, Robbins JA, Roecker EB, Coyle JL, Wood JL. A penetration-aspiration scale. Dysphagia. 1996 Spring;11(2):93-8. doi: 10.1007/BF00417897. PMID 8721066

RESULTS

PARTICIPANT FLOW:
Groups:
- Amyotrophic Lateral Sclerosis (ALS): Adults with a neurologist-confirmed diagnosis of ALS who completed a videofluoroscopy involving swallows of different liquid consistencies.
- Parkinson Disease: Adults with a neurologist-confirmed diagnosis of Parkinson Disease who completed a videofluoroscopy involving swallowing of different consistencies of liquid.
Period: Overall Study
Arm/Group | Amyotrophic Lateral Sclerosis (ALS) | Parkinson Disease
Started | 20 | 20
Completed | 20 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Amyotrophic Lateral Sclerosis: We will be recruiting individuals with confirmed or probably ALS, who experience speech or swallowing problems, to attend one data collection session. All participants will undergo the same protocol, including a Videofluoroscopic Swallowing Examination, and Tongue Strength Measurement.
  Videofluoroscopic Swallowing Examination: During the videofluoroscopy, subjects will take up to 21 sips of liquid, ranging in thickness from thin (like water), to extremely-thick (like pudding or custard). The liquids will be mixed with E-Z-Paque barium sulfate, to allow it to be visible on the x-ray.
  Tongue Strength Measurement: We will measure tongue strength using a tongue pressure measurement system called the Iowa Oral Performance Instrument (IOPI). A small disposable bulb filled with air will be placed in the mouth, just behind the front teeth. Participants will be asked to press their tongue upwards against the bulb as hard as they can, three (3) times at the front of the tongue and three (3) times at the back of the tongue (i.e., total of six (6) maximum isometric tongue presses). Participants will also be asked to swallow their saliva with the bulb placed in their mouth, three (3) times.
  Tongue pressure measurement will be completed twice in the data collection session - once at the beginning, and once at the end (following the videofluoroscopy).
- Parkinson's Disease: We will be recruiting individuals with a diagnosis of Parkinson's disease, who experience speech or swallowing problems, to attend one data collection session. All participants will undergo the same protocol, including a Videofluoroscopic Swallowing Examination, and Tongue Strength Measurement.
  Videofluoroscopic Swallowing Examination: During the videofluoroscopy, subjects will take up to 21 sips of liquid, ranging in thickness from thin (like water), to extremely-thick (like pudding or custard). The liquids will be mixed with E-Z-Paque barium sulfate, to allow it to be visible on the x-ray.
  Tongue Strength Measurement: We will measure tongue strength using a tongue pressure measurement system called the Iowa Oral Performance Instrument (IOPI). A small disposable bulb filled with air will be placed in the mouth, just behind the front teeth. Participants will be asked to press their tongue upwards against the bulb as hard as they can, three (3) times at the front of the tongue and three (3) times at the back of the tongue (i.e., total of six (6) maximum isometric tongue presses). Participants will also be asked to swallow their saliva with the bulb placed in their mouth, three (3) times.
  Tongue pressure measurement will be completed twice in the data collection session - once at the beginning, and once at the end (following the videofluoroscopy).
- Total: Total of all reporting groups
Arm/Group | Amyotrophic Lateral Sclerosis | Parkinson's Disease | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 65 [53 to 70] | 70 [65 to 75] | 67 [58 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 4 | 14
  Male | 10 | 16 | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 19 | 19 | 38
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 18 | 19 | 37
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 20 | 20 | 40

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Residue of Concern (Observational)
Description: Residue is material remaining behind in the pharynx after the swallow. We measured residue by tracing the area of barium visible on a lateral view x-ray (in pixels, using ImageJ software) and dividing that area by the squared length C2-C4 cervical spine. This cervical spine scalar provides a common anatomical reference that is a proxy for pharyngeal size, and enables the comparison of residue severity across different people with different neck length and pharynx size. Smaller values are considered better. The 75th percentile healthy reference values for this measure are 1.7% on thin liquids, 1.9% on slightly thick liquids, 2.2% on mildly thick liquids, 1.6% on moderately thick liquids and 1.5% on extremely thick liquids. Values above these thresholds are considered atypical and of clinical concern. We report the number of participants who display atypical total pharyngeal residue measures per consistency.
Time Frame: Single timeframe (baseline only)
Population: Two cohorts of participants were enrolled in this observational study: 1) A cohort of 20 adults with Amyotrophic Lateral Sclerosis (ALS); and 2) A cohort of 20 adults with Parkinson disease. Due to data quality issues, partial data were missing for some consistencies.
Measure: Count of Participants; unit: Participants
Groups:
- Amyotrophic Lateral Sclerosis: Thin Liquids; Parkinson Disease: Thin Liquid: Participants were asked to swallow a series of 3 comfortably sized sips of thin liquid barium (Bracco E-Z-Paque powder prepared in 20% w/v concentration with water) and swallow when ready (without a cue).
- Amyotrophic Lateral Sclerosis: Slightly Thick Liquids; Parkinson Disease: Slightly Thick Liquids: Participants were asked to swallow a series of 3 comfortably sized sips of slightly thick liquid barium (Bracco E-Z-Paque powder prepared in 20% w/v concentration with water and Nestle Resource Thicken Up Clear Xanthan Gum thickener) and swallow when ready (without a cue).
- Amyotrophic Lateral Sclerosis: Mildly Thick Liquids; Parkinson Disease: Mildly Thick Liquids: Participants were asked to swallow a series of 3 comfortably sized sips of mildly thick liquid barium (Bracco E-Z-Paque powder prepared in 20% w/v concentration with water and Nestle Resource Thicken Up Clear Xanthan Gum thickener) and swallow when ready (without a cue).
- Amyotrophic Lateral Sclerosis: Moderately Thick Liquids; Parkinson Disease: Moderately Thick Liquids: Participants were asked to swallow a series of 3 comfortably sized sips of moderately thick liquid barium (Bracco E-Z-Paque powder prepared in 20% w/v concentration with water and Nestle Resource Thicken Up Clear Xanthan Gum thickener) and swallow when ready (without a cue).
- Amyotrophic Lateral Sclerosis: Extremely Thick Liquids; Parkinson Disease: Extremely Thick Liquids: Participants were asked to swallow a series of 3 comfortably sized sips of extremely thick liquid barium (Bracco E-Z-Paque powder prepared in 20% w/v concentration with water and Nestle Resource Thicken Up Clear Xanthan Gum thickener) and swallow when ready (without a cue).
Arm/Group | Amyotrophic Lateral Sclerosis: Thin Liquids | Amyotrophic Lateral Sclerosis: Slightly Thick Liquids | Amyotrophic Lateral Sclerosis: Mildly Thick Liquids | Amyotrophic Lateral Sclerosis: Moderately Thick Liquids | Amyotrophic Lateral Sclerosis: Extremely Thick Liquids | Parkinson Disease: Thin Liquid | Parkinson Disease: Slightly Thick Liquids | Parkinson Disease: Mildly Thick Liquids | Parkinson Disease: Moderately Thick Liquids | Parkinson Disease: Extremely Thick Liquids
Number analyzed (Participants) | 20 | 19 | 18 | 17 | 17 | 17 | 17 | 17 | 17 | 17
Participants | 6 | 6 | 3 | 6 | 4 | 2 | 3 | 3 | 1 | 2

2. Primary Outcome: Maximum Anterior Isometric Tongue Pressure
Description: Tongue strength was measured using a tongue pressure measurement system called the Iowa Oral Performance Instrument (IOPI). A small disposable bulb filled with air was placed in the mouth, just behind the front teeth. Participants were asked to press the front of their tongue upwards against the bulb as hard as possible. This task was repeated 3 times. The maximum value obtained across 3 repetitions was recorded as "maximum anterior isometric pressure". Higher values represent greater tongue strength. We report group mean values and standard deviations for this measure.
Time Frame: Single timeframe (baseline only)
Population: Two cohorts of participants were enrolled: 1) A cohort of 20 adults with Amyotrophic Lateral Sclerosis (ALS); and 2) A cohort of 20 adults with Parkinson disease. Due to data quality issues, anterior isometric pressure data were missing for 3 of the participants with ALS.
Measure: Mean (Standard Deviation); unit: kilopascals
Groups:
- Amyotrophic Lateral Sclerosis: Individuals with a neurologist-confirmed diagnosis of ALS.
- Parkinson Disease: Individuals with a neurologist-confirmed diagnosis of Parkinson Disease.
Arm/Group | Amyotrophic Lateral Sclerosis | Parkinson Disease
Number analyzed (Participants) | 17 | 20
kilopascals | 34 (19) | 55 (17)
Statistical Analysis 1: Comparison: Amyotrophic Lateral Sclerosis vs Parkinson Disease; This was an observational study. The statistical test explores whether there were significant differences in tongue pressure between the two cohorts. The hypothesis was that individuals with ALS would display significantly lower maximum anterior isometric tongue pressures compared to the people with PD; Test type: Superiority; p < 0.001, ANOVA — A priori threshold for statistical significance was p < 0.05; Cohen's d = 1.18 — Cohen's d values > 0.8 are considered large

3. Primary Outcome: Regular Effort Saliva Swallow Tongue Pressure
Description: Tongue strength was measured using a tongue pressure measurement system called the Iowa Oral Performance Instrument (IOPI). A small disposable bulb filled with air was placed in the mouth, just behind the front teeth. Participants were asked to swallow their saliva with the bulb in this position. This task was repeated 3 times. The mean value obtained across 3 repetitions was recorded as "regular effort saliva swallow tongue pressure". Higher values represent greater tongue strength. We report group mean values and standard deviations for this measure.
Time Frame: Single timeframe (baseline only)
Population: Two cohorts of participants were enrolled: 1) A cohort of 20 adults with Amyotrophic Lateral Sclerosis (ALS); and 2) A cohort of 20 adults with Parkinson disease. Due to data quality issues, saliva swallow tongue pressure data were missing for 3 of the participants with ALS.
Measure: Mean (Standard Deviation); unit: kilopascals
Groups:
- Amyotrophic Lateral Sclerosis: We will be recruiting individuals with confirmed or probably ALS, who experience speech or swallowing problems, to attend one data collection session.
  Tongue Strength Measurement: We will measure tongue strength using a tongue pressure measurement system called the Iowa Oral Performance Instrument (IOPI). A small disposable bulb filled with air will be placed in the mouth, just behind the front teeth. Participants will be asked to press their tongue upwards against the bulb as hard as they can, three (3) times at the front of the tongue and three (3) times at the back of the tongue (i.e., total of six (6) maximum isometric tongue presses). Participants will also be asked to swallow their saliva with the bulb placed in their mouth, three (3) times.
- Parkinson's Disease: We will be recruiting individuals with a diagnosis of Parkinson's disease, who experience speech or swallowing problems, to attend one data collection session.
  Tongue Strength Measurement: We will measure tongue strength using a tongue pressure measurement system called the Iowa Oral Performance Instrument (IOPI). A small disposable bulb filled with air will be placed in the mouth, just behind the front teeth. Participants will be asked to press their tongue upwards against the bulb as hard as they can, three (3) times at the front of the tongue and three (3) times at the back of the tongue (i.e., total of six (6) maximum isometric tongue presses). Participants will also be asked to swallow their saliva with the bulb placed in their mouth, three (3) times.
Arm/Group | Amyotrophic Lateral Sclerosis | Parkinson's Disease
Number analyzed (Participants) | 17 | 20
kilopascals | 19 (12) | 17 (8)
Statistical Analysis 1: Comparison: Amyotrophic Lateral Sclerosis vs Parkinson's Disease; This was an observational study rather than a trial. The hypothesis was that individuals with ALS would display significantly lower regular effort saliva swallow pressures than the individuals with PD; Test type: Superiority; p < 0.001, ANOVA; Cohen's d = 1.75 — Cohen's d values > 0.8 are considered large

4. Primary Outcome: Number of Participants With Unsafe Swallows (Observational)
Description: Swallowing safety was measured using the 8-point Penetration-Aspiration Scale, an 8-point categorical scale which captures the depth to which any material enters the airway and whether or not the material is ejected. Levels 1 and 2 on the scale are considered safe, while levels > 2 are considered unsafe. Actual scale scores (1-8) were recorded and then converted to binary categorical scores (< 3 vs >/= 3). We report the frequency (count) of participants showing scores > 2 by bolus consistency.
Time Frame: Baseline (Single timepoint only)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Amyotrophic Lateral Sclerosis: Thin Liquids | Amyotrophic Lateral Sclerosis: Slightly Thick Liquids | Amyotrophic Lateral Sclerosis: Mildly Thick Liquids | Amyotrophic Lateral Sclerosis: Moderately Thick Liquids | Amyotrophic Lateral Sclerosis: Extremely Thick Liquids | Parkinson Disease: Thin Liquid | Parkinson Disease: Slightly Thick Liquids | Parkinson Disease: Mildly Thick Liquids | Parkinson Disease: Moderately Thick Liquids | Parkinson Disease: Extremely Thick Liquids
Number analyzed (Participants) | 20 | 19 | 18 | 17 | 17 | 17 | 17 | 17 | 17 | 17
Participants | 10 | 9 | 7 | 6 | 3 | 2 | 1 | 1 | 0 | 1

5. Secondary Outcome: Maximum Posterior Isometric Tongue Pressure (Observational).
Description: Tongue strength was measured using a tongue pressure measurement system called the Iowa Oral Performance Instrument (IOPI). A small disposable bulb filled with air was placed in the mouth, with the front margin of the sensor aligned with the first molar tooth. Participants were asked to press the back of their tongue upwards against the bulb as hard as possible. This task was repeated 3 times. The maximum value obtained across 3 repetitions was recorded as "maximum posterior isometric pressure". Higher values represent greater tongue strength. We report group mean values and standard deviations for this measure. There was no statistical analysis comparing group values for this parameter.
Time Frame: Single timeframe (baseline only)
Population: Two cohorts of participants were enrolled: 1) A cohort of 20 adults with Amyotrophic Lateral Sclerosis (ALS); and 2) A cohort of 20 adults with Parkinson disease. Due to data quality issues, posterior isometric pressure data were missing for 3 of the participants with ALS.
Measure: Mean (Standard Deviation); unit: kilopascals
Arm/Group | Amyotrophic Lateral Sclerosis | Parkinson Disease
Number analyzed (Participants) | 17 | 20
kilopascals | 29 (20) | 51 (19)

6. Secondary Outcome: Number of Participants With Multiple Swallows Per Bolus (Observational)
Description: The number of swallows needed to clear a single bolus will be counted. A single swallow is considered efficient, while 2+ swallows for one bolus is considered atypical. We will report the number of participants with > 1 swallow per bolus.
Time Frame: Single timeframe (baseline only)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Amyotrophic Lateral Sclerosis: Thin Liquids | Amyotrophic Lateral Sclerosis: Slightly Thick Liquids | Amyotrophic Lateral Sclerosis: Mildly Thick Liquids | Amyotrophic Lateral Sclerosis: Moderately Thick Liquids | Amyotrophic Lateral Sclerosis: Extremely Thick Liquids | Parkinson Disease: Thin Liquid | Parkinson Disease: Slightly Thick Liquids | Parkinson Disease: Mildly Thick Liquids | Parkinson Disease: Moderately Thick Liquids | Parkinson Disease: Extremely Thick Liquids
Number analyzed (Participants) | 20 | 19 | 18 | 17 | 17 | 17 | 17 | 17 | 17 | 17
Participants | 6 | 8 | 9 | 5 | 8 | 6 | 3 | 2 | 2 | 2

7. Secondary Outcome: Number of Participants Displaying Prolonged Pharyngeal Bolus Transit (Observational)
Description: The time interval from the first frame showing the bolus entering the pharynx (passing the shadow of the ramus of the mandible) until the first frame showing the bolus entering the upper esophageal sphincter was calculated (in milliseconds) for each bolus. The 75th percentile healthy reference values for this measure are 533 ms on thin liquids, 567 ms on slightly thick liquids, 701 ms on mildly thick liquids, 867 ms on moderately thick liquids and 1001 ms on extremely thick liquids. Pharyngeal transit durations above these values are considered prolonged and atypical. We will report the number of participants who present with atypical pharyngeal transit duration above these 75th percentile reference value thresholds per consistency.
Time Frame: Single timeframe (baseline only)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Amyotrophic Lateral Sclerosis: Thin Liquids | Amyotrophic Lateral Sclerosis: Slightly Thick Liquids | Amyotrophic Lateral Sclerosis: Mildly Thick Liquids | Amyotrophic Lateral Sclerosis: Moderately Thick Liquids | Amyotrophic Lateral Sclerosis: Extremely Thick Liquids | Parkinson Disease: Thin Liquid | Parkinson Disease: Slightly Thick Liquids | Parkinson Disease: Mildly Thick Liquids | Parkinson Disease: Moderately Thick Liquids | Parkinson Disease: Extremely Thick Liquids
Number analyzed (Participants) | 18 | 19 | 17 | 15 | 17 | 17 | 17 | 17 | 17 | 17
Participants | 5 | 10 | 7 | 7 | 8 | 5 | 4 | 5 | 5 | 6

ADVERSE EVENTS:
Time Frame: 1 week following the single appointment data collection session
Description: Standard definitions were used
Arm/Group | Amyotrophic Lateral Sclerosis | Parkinson's Disease
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20

LIMITATIONS AND CAVEATS:
This was an observational study. For the majority of measures, we report count data for each cohort but do not compare frequencies across cohorts or across conditions (i.e. bolus consistencies) within cohort.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-10-19): https://cdn.clinicaltrials.gov/large-docs/58/NCT03192358/Prot_SAP_000.pdf